CLINICAL TRIAL: NCT05075473
Title: SEGMENTAL STABILIZATION AND GENERAL LUMBER STABILIZATION EXERCISE IN CHRONIC LOW BACK PAIN
Brief Title: SEGMENTAL AND GENERAL STABILIZATION EXERCISES IN CHRONIC LOW BACK PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1703-MPHIL-OPT/008
Record Dates: First submitted 2020-04-09; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2020-04

CONDITIONS: Segmental Stabilization; Generalized Segmental Stabilization Exercises

STUDY DESIGN:
Intervention Model Description: 44 patients with chronic low back pain, distributed randomly in to two groups.
Who Masked: Investigator
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmental Stabilization (Experimental): Segmental control over the primary stabilizers (TrA, deep multifidus, pelvic floor and diaphram) is maintained. Weight of body is minimized by using drawing in maneuver. Time duration will be of 30 to 40 mins, thrice a week for four weeks. Hot packs will be applied for 10 mins. In starting days, 8 to 10 reps with hold time 5 count. In later days, 12 to 15 reps with hold time increases up till 10 to 15 counts.
  Interventions: Other: Segmental stabilization
- General lumber stabilization exercises (Active Comparator): It includes exercises in closed chain with low velocity as well as low load. Time duration will be of 30 to 40 mins, thrice a week for four weeks. Hot packs will be applied for about 10 mins. In starting days, 8 to 10 reps with hold time 5 count. In later days, 12 to 15 reps with hold time increases up till 10 to 15 counts.
  Interventions: Other: Generalized Lumber stabilization exercsies

INTERVENTIONS:
Other: Segmental stabilization — Physiotherapist will perform activation of multifidus in prone position. It also includes activation of transverse abdominas in crook lying position, in sitting as well as in point kneeling position to re-establish simultaneous contraction of deep muscles synergy.
  Other Names: Experimental
  Arms: Segmental Stabilization
Other: Generalized Lumber stabilization exercsies — It can by performed by patient him or her self under physiotherapist's assistance. Lumber neutral position is maintained. Bridging in prone as well as supine position will be maintained.
  Other Names: Active comparator
  Arms: General lumber stabilization exercises

SUMMARY:
Chronic low back pain effects more than 50% of general population. It's prevalence is higher is young adults that are economically active adults.

Its significance is often underestimated because usually young adults ignore these initial episodes of low back pain due to their busy life style or life full of commitments. Approximately 70% of adults have at least one episode of low back pain during their lifetimes.

DETAILED DESCRIPTION:
It will be randomized control trial with 60 patients with chronic low back pain divided into 2 groups. One group will be given segmental stabilization whose purpose is to achieve segmental control over primary stabilizers. Second group will be given just generalized lumber stabilization exercises as it includes close chain exercises with low velocity as well as low load. This study will be conducted in Rehabilitation setup of Benazir Bhutto hospital Rawalpindi and IIRS that is Rehabilitation dept. at Al Nafees medical college and hospital, Islamabad. Non probability Convenience Sampling technique will be utilized

ELIGIBILITY:
Inclusion Criteria:

* Both males and females will be included in the study

Exclusion Criteria:

* Age limits of subjects will be between 15 to 60

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
VAS | 4 weeks (1st reading is at the baseline, 2nd is at 3rd day, 3rd is at 5th day, 4th is at 8th day, 5th is at 10th day, 6th is at 12th day, 7th is at 19th day and 8th reading is at 26th day.
  Visual analogue scale for Pain 0= no pain, 10= unbearable pain
Oswestry disability Index | 4 weeks (1st reading is at the baseline, 2nd is at 3rd day, 3rd is at 5th day, 4th is at 8th day, 5th is at 10th day, 6th is at 12th day, 7th is at 19th day and 8th reading is at 26th day.
  It is used to measure permanent functional disability. For each section, total possible score is 5, after completing all 10 sections. sum of all scores will be obtained in the form of percentages.
International physical activity questionnaire | Only one reading is required that is the baseline reading.
  It is used to measure to physical activity of a person

OTHER OUTCOMES:
ROM | 4 weeks (1st reading is at the baseline, 2nd is at 3rd day, 3rd is at 5th day, 4th is at 8th day, 5th is at 10th day, 6th is at 12th day, 7th is at 19th day and 8th reading is at 26th day.
  It is an acronym of Range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Summaiya Zaman, Mphil, Principal Investigator — Isra Institute of rehabilitation
Locations (1):
- Isra institute of rehabilitation sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No